CLINICAL TRIAL: NCT02566967
Title: An Evaluation of the Optimal Dose of Tofacitinib Needed to Achieve LDA or Clinical Remission in Patients With Active Rheumatoid Arthritis (RA) as Measured From a Clinical and Structural Perspective When Treating to Target
Brief Title: An Evaluation of the Optimal Dose of Tofacitinib Needed to Achieve Low Disease Activity (LDA) or Clinical Remission in Patients With Active Rheumatoid Arthritis (RA) as Measured From a Clinical and Structural Perspective
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norman B. Gaylis, MD (Other)
Responsible Party: Sponsor-Investigator, Norman B. Gaylis, MD, MD, Arthritis & Rheumatic Disease Specialties Research
Organization: Arthritis & Rheumatic Disease Specialties Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-012015
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Other): open label use of tofacitinib at either 5 mg bid or 10 mg bid delending on treat to target goal
  Interventions: Drug: tofacitinib

INTERVENTIONS:
Drug: tofacitinib — oral tofacitinib will be taken 2 times daily

SUMMARY:
This study will evaluate the optimal dose of tofacitinib needed to achieve low disease activity (LDA) or clinical remission as measured by the CDAI score. Once LDA or clinical remission has been achieved, the structural benefit in reducing erosions, synovitis and bone edema as measured by low field MRI will be determined at the same time period by the use of the OMERACT/RAMRIS scoring system

DETAILED DESCRIPTION:
This study will evaluate the optimal dose of tofacitinib needed to achieve low disease activity (LDA) or clinical remission as measured by the CDAI score. Once LDA or clinical remission has been achieved, the structural benefit in reducing erosions, synovitis and bone edema as measured by low field MRI will be determined at the same time period by the use of the OMERACT/RAMRIS scoring system and correlated to the clinical findings. The target for each patient will be determined at the time of study entry depending on the degree of disease activity of the individual patient. This is based on the understanding that LDA is an acceptable goal in certain patients with long standing disease or high disease activity. If the patient reaches LDA while taking tofacitinib at a 5 mg b.i.d. dose, the patient will be given the opportunity to have the dose increased to 10 mg b.i.d. in the hopes of reaching clinical remission.

There are two treat to target goals: Clinical Remission as defined by a CDAI score of <2.8 for those patients who entered the study with a CDAI score of <22 and Low Disease Activity (LDA) as defined by a CDAI score of <10 for those who entered the study with a CDAI score of > 22.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years old at the screening visit
2. Patient must be able to understand the information provided to them and give written Informed Consent
3. Female subjects of childbearing potential must test negative for pregnancy
4. Male and female subjects of childbearing potential must agree to use two highly effective methods of contraception throughout the study and for at least 3 months after the last dose of tofacitinib.
5. Female patients who are not of childbearing potential must either be postmenopausal for at least 12 months or have undergone a documented hysterectomy and/or bilateral oophorectomy.
6. Patients can be naïve to biologic therapy or have had exposure to TNF or biologic therapy (see appropriate wash out schedule) and be experiencing at least a moderate disease activity score as determined by a CDAI of > 10 at Screening despite currently receiving Methotrexate therapy at a dose of 10-25 mg/weekly for at least 12 weeks and at a stable dose for the past 4 weeks.
7. Patients on prednisone must be receiving a daily dose of < 10 mg.
8. Subjects must screen negative for active tuberculosis (TB) by either a PPD or a QuantiFERON Gold test (unless previously performed and documented within 3 months prior to screening). If patient tests positive for latent TB at screening, the chest X-ray at Screening must be negative for active TB and the patient must be started on ( or have completed) an adequate course of therapy for latent tuberculosis at the Baseline visit. Patient must complete the entire 9 month course of treatment for latent TB.
9. Chest radiograph taken at screening (unless taken and documented within 3 months prior to screening) must be negative for active TB and have non clinically significant medical findings.
10. Patients must be able and willing to comply with the requirements of the study protocol

Exclusion Criteria:

1. Patients who have a history of any inflammatory disease which would be interfere with outcome measurement
2. Patients who in the Investigator's opinion have a medical condition in which participation in this trial is contraindicated
3. Patients who have received intramuscular, intravenous, or intraarticular (IM/IV/IA) corticosteroids 28 days prior to baseline.
4. Patients who have active TB or a history of active TB (positive PPD skin test >5mm and a positive chest x-Ray) or patients who have come in close contact with an individual with active TB.
5. Patients with a history of acute or chronic viral hepatitis B or C or those who test positive at screening.
6. Patients with a known human immunodeficiency virus (HIV) infection.
7. Concurrent malignancy or a history of malignancy other than a non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
8. Patients who have a metal device affected by MRI (e.g. any type of electronic, mechanical or magnetic implant; cardiac pacemaker; aneurysm clip(s); implanted cardioverter defibrillator; or cochlear implant)
9. Patients who have potential ferromagnetic foreign body (metal slivers metal shavings, other metal objects) for which they have sought medical attention
10. Patients at a high risk of infection in the Investigator's opinion or have had recurrent infections requiring hospitalization or parenteral antimicrobial therapy within the past 6 months.
11. Patients with an adverse reaction to tofacitinib
12. Patients with any other condition (e.g., clinically significant laboratory values) which in the Investigator's judgment would make the patient unsuitable for inclusion in this study
13. Patients who have received prohibited medications:

the following approved biological therapy for RA: etanercept, adalimumab, anakinra, abatacept, tocilizumab within 28 days of baseline

* rituximab within 9 months of baseline
* infliximab within 56 days of baseline
* DMARDs other than methotrexate within 28 days of baseline
* any experimental biologic agent within three months or 5 half-lives prior to baseline
* exposure to JAK inhibitor 14. Female patients who are breast-feeding, pregnant, or plan to become pregnant during the trial or within twelve weeks following last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Record the optimal dose of tofacitinib needed to achieve LDA or clinical remission as measured by CDAI score | one year
  the daily dosed used in patients to achieve LDA

SECONDARY OUTCOMES:
low -field (0.3T) MRI will be used to measure the reduction of synovitis and bone edema | one year
  was synovitis, bone edema and erosion reduced
correlation of the structural and clinical responses performed the structural outcomes as measured by MERERACT and correlate them to the clinical responses and dose adjustments made during the course of the study | one year
  was there a correlation is structural and clinical response
record the number of patients who reach low disease activity and a measurable structural response | one year
  the number of patient who reached LDA and a measurable structural change
record the number of patients in which structural response occurred without clinical response | one year
  number of patients who had a structural response but no clinical response
record the number of patients who required an increase in the dose of tofacitinib due to lack of clinical response from Baseline as measured by CDAI score | one year
  number of patients who had dose escalated to 10 mg bid
record the change in CDAI score for all patients from Baseline through the last dose of the initial dose (5 mg b.i.d) of tofacitinib | one year
  record CDAI scores from Baseline to Week 52
record the change in CDAI score from the step up period ( 10 mg b.i.d) to the end of the dosing period | one year
  record CDAI score at dose 10 mg bid

CONTACTS AND LOCATIONS:
Locations (1):
- AARDS Research, Inc., Aventura, Florida, United States